CLINICAL TRIAL: NCT04515511
Title: Medical Intensive Care Unit of PUMCH
Brief Title: Whether a Minimal Volume Could Predict Fluid Responsiveness Using Thermodilution by PAC in Septic Shock Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH fc
Record Dates: First submitted 2020-08-10; First posted 2020-08-17 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Septic Shock; Hemodynamic Instability; Fluid Therapy
Keywords: Sepsis/Septic shock; Hemodynamic monitor; Fluid challenge; Cardiac output; Pulmonary artery catheter; Thermodilution
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Gelatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- standard care (Experimental): ICU septic shock patients with refractory hypotension with indwelling pulmonary artery catheter received five sequential intravenous boluses of 100 mL 4% gelatin. Cardiac output measured by thermodilution of PAC before fluid challenge (baseline) and three minutes after each bolus. Fluid responsiveness (FR) was defined as an increase in CO greater than 10% after 500 mL fluid infusion. The smallest volume which can perform an effective fluid challenge was analyzed.
  Interventions: Other: 4% gelatin

INTERVENTIONS:
Other: 4% gelatin — Pulmonary artery catheter insertion is prepared before fluid challenge. Baseline hemodynamic value and each time after 5 sequential intravenous boluses of 100 mL colloid are recorded.
  Other Names: Pulmonary artery catheter

SUMMARY:
Assessment of fluid responsiveness (FR) is to detect whether patient could benefit from fluid therapy. Mini fluid challenge has been widely used in clinical practice to prevent patients from volume overload. In clinical practice, 100 mL or 250 mL have been used most frequently and FR was defined as an increase in CO greater than 10% as much as the changes in CO after infusion of 500 mL. While using a half of volume infusion and assessed by the traditional standard of FR, this might misclassify more patients as nonresponders. In that it is imperative to test the predictive ability of mini fluid and find out the threshold of cutoff value. Meanwhile, in almost mini-FC, cardiac output were measured by echocardiography(VTi) and pulse contour,None of the studies conducted cardiac output (CO)measurement by gold standard method of thermodilution by pulmonary artery catheter (PAC). The correlation between new generated CO measurements and PAC varies in different studies as well. It is imperative to investigate the reliability of mini-FC to predicting fluid responsiveness(FR).The investigator's study is to detect the predictive minimal volume using thermodilution by PAC in septic shock patient.

DETAILED DESCRIPTION:
Fluid therapy is the cornerstone of septic resuscitation. In recent decade, a restrictive fluid strategy has been applied to shock resuscitation for fewer complications and shorter hospital stays compared with a liberal fluid strategy. Therefore, it is a reasonable step to assess the patient's response to fluid infusion to avoid excessive fluid administration.Mini-fluid challenge allows the selection of fluid responders by inducible changes of hemodynamic parameters after changing the preload gaining popularity. The mini fluid challenge was firstly described by Muller et al. in 2011. They found an infusion of 100 mL colloid over 1 minute and the assessment by cardiac output using velocity time integral (VTi) at the aortic outflow tract could predict fluid responsiveness (FR). Since then, a total of seven investigations have been published. Although a mini-fluid challenge may help the decision-making process of fluid management, the investigation results differed from each other, especially in minimal volume and cut off value of hemodynamic parameters change. Meanwhile, we noticed that when measuring CO, the method of thermodilution by pulmonary artery catheter (PAC), which is the gold standard of CO measurement, was not used in these studies. Furthermore, the majority participants of the studies were perioperative patients in a stable hemodynamic state.Therefore, there are two question needed to be answered:what is the minimal infusion volume in effectively predicting fluid responsiveness, and whether mini-volume can perform a real change in septic shock patients. Thus, it is necessary to explore the minimal volume in fluid challenge by PAC and test its reliability in detecting responders (R) and nonresponders (NR).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosis of septic shock and is required fluid challenge in the presence of invasive hemodynamic monitoring.
* Patients with hypotension (SBP <90 mmHg or MAP <65 mmHg)
* Patients with evidences of tissue hypoperfusion (including but not limited to oliguria, skin mottling, altered mental status, cool peripheries, hyperlactatemia, et al).

Exclusion Criteria:

* Age less than 18yrs or greater than 80yrs
* Shock is diagnosed with other types of shock
* Known allergy to colloid fluids
* Pregnancy
* Recent participation in another biomedical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | Baseline and immediately after each bolus of 100 mL colloid, average 3 minutes
  Cardiac output measured by therm-dilution of pulmonary artery catheter. An increase in cardiac output(CO) greater than 10% after a volume expansion of 500 mL is defined as fluid responsiveness(FR).

SECONDARY OUTCOMES:
Oxygen saturation | Baseline and immediately after each bolus of 100 mL colloid, average 3 minutes
  Oxygen saturation can be obtained directly from blood gas include which reflects extraction of oxygen and assess whether CO is sufficient enough to meet patient's enough.
Carbon dioxide partial pressure | Baseline and immediately after each bolus of 100 mL colloid, average 3 minutes
  PCO2 can be obtained directly from blood gas. It is considered as alternative markers of tissue hypoperfusion and attempted to be used to guide treatment for shock.
Hemoglobin | Baseline and immediately after each bolus of 100 mL colloid, average 3 minutes
  Hemoglobin will be diluted during fluid challenge and it is also an important index to guide fluid resuscitation by improving extraction of oxygen and optimizing oxygen delivery.
Heart rate | Baseline and immediately after each bolus of 100 mL colloid, average 1 minutes
  Heart rate is monitored to assess the effect of the fluid challenge
Mean arterial pressure | Baseline and immediately after each bolus of 100 mL colloid, average 1 minutes
  Mean arterial pressure is monitored to assess the effect of the fluid challenge
Central venous pressure | Baseline and immediately after each bolus of 100 mL colloid, average 1 minutes
  Central venous pressure is monitored to assess the preload status and effect of the fluid challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Li Weng, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
In our department, we has done a serial clinical studies of fluid challenge, we will do retrospective study first.

REFERENCES:
- [Derived] Yang T, Weng L, Jiang W, Li S, Du B. Hemodynamic effects of different fluid volumes for a fluid challenge in septic shock patients. Chin Med J (Engl). 2022 Mar 20;135(6):672-680. doi: 10.1097/CM9.0000000000001919. PMID 34935687